CLINICAL TRIAL: NCT00395603
Title: Compare Ezetimibe 10mg and Simvastatin 40mg vs Atorvastatin 80mg Daily in Subjects With Cardiovascular Heart Disease and/or Diabetes Mellitus With Uncontrolled Lipids on Statin Therapy
Brief Title: Vytorin Treating Uncontrolled Lipids (VyTUL) Study (0653A-122)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated early due to poor recruitment.
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0653A-122; 2006_042
Record Dates: First submitted 2006-11-02; First posted 2006-11-03 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus | interventions — Ezetimibe; Simvastatin; Duration of Therapy

INTERVENTIONS:
Drug: MK0653A, ezetimibe (+) simvastatin / Duration of Treatment: 6 Weeks
Drug: Comparator: atorvastatin / Duration of Treatment: 6 Weeks

SUMMARY:
To compare the effectiveness of ezetimibe/simvastatin 10/40 daily to atorvastatin 80 daily in reducing the concentration of ldl-c at endpoint after 6 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age
* Treated for at least the last 3 months with a daily dose of atorvastatin 40 mg
* Existing coronary heart disease and cholesterol > 4.0 mmol/l

Exclusion Criteria:

* Uncontrolled diabetes
* Elevated liver function tests
* Elevated creatine kinase (ck)
* Triglycerides (tg) > 4.5 mmol/l
* Drug or alcohol dependency within 6 months prior to visit 1
* Woman receiving hormonal therapy who have not been maintained on a stable dose and regimen for at least 8 weeks and are willing to continue the same regimen for the duration of the study
* Woman of childbearing potential not using an acceptable method of birth control
* Women who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2006-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Percentage reduction in ldl-c at end-point after 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC